CLINICAL TRIAL: NCT01875718
Title: A Randomized, Double-blind, Placebo-controlled Parallel-group Study on Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of UC1010 Administered Subcutaneously, Single-dosing in Healthy Women (Part 1) and Multiple Dosing in PMDD Women (Part 2) - Phase I/II Study
Brief Title: A Phase I/II Study to Evaluate UC1010 Treatment in Premenstrual Dysphoric Disorder (PMDD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Umecrine Mood AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UM104
Record Dates: First submitted 2013-05-29; First posted 2013-06-12 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Premenstrual Dysphoric Disorder
MeSH Terms: conditions — Premenstrual Dysphoric Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- UC1010 low dose (Active Comparator)
  Interventions: Drug: UC1010
- UC1010 high dose (Active Comparator)
  Interventions: Drug: UC1010
- Vehicle (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UC1010
  Arms: UC1010 high dose; UC1010 low dose
Drug: Placebo
  Arms: Vehicle

SUMMARY:
The study is a phase 1/2 study in two parts. In part 1, the primary objective is to assess the pharmacokinetics of UC1010 when administered subcutaneously as a single dose to healthy women. The safety and tolerability of UC1010 is also evaluated in study part 1.

In part 2, the primary objective is to assess the pharmacodynamic effect of UC1010 on premenstrual symptoms in women with Premenstrual Dysphoric Disorder (PMDD) when given during the luteal phase of the menstrual cycle. The pharmacodynamic effect is evaluated through the patients' daily ratings of premenstrual symptoms. In both study parts, two active treatment groups are compared to one placebo group.

ELIGIBILITY:
Inclusion Criteria:

Part 1 -Essentially healthy

Part 2 -Have PMDD according to DSM-IV verified in two menstrual cycles

Exclusion Criteria:

* steroid hormonal treatment during the previous three months
* treatment with psychopharmaceuticals or other treatment for PMS
* history of or a significant medical condition ongoing
* be pregnant or plan a pregnancy within the study period

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Premenstrual symptom severity | Daily Record of Severity of Problems (DRSP) measured during 4-5 months

SECONDARY OUTCOMES:
Number of subjects with adverse events | During 1.5 month (starting from first dose)

CONTACTS AND LOCATIONS:
Locations (1):
- Umecrine Mood AB, Solna, Sweden